CLINICAL TRIAL: NCT01349842
Title: CirCe01 Study: Evaluation of the Use of Circulating Tumour Cells to Guide Chemotherapy From the 3rd Line of Chemotherapy for Metastatic Breast Cancer
Brief Title: Circulating Tumor Cells to Guide Chemotherapy for Metastatic Breast Cancer
Acronym: CirCé01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2009-03
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Ductal Infiltrating Metastatic
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Circulating Tumor Cells (Experimental): Centralized determination of CTC by CellSearch® technology (Veridex), the only technology currently validated in clinical practice for the early evaluation of response to chemotherapy of breast cancers. This evaluation is performed by blood sampling comparing the CTC level before the first injection of each new line of chemotherapy. Chemotherapy can only be continued in the case of a positive CTC response. Discontinuation of chemotherapy can also be decided by the clinician on the basis of other clinical or radiological arguments.
  Interventions: Biological: Blood sampling
- Clinical and radiological criteria (Other): Management of chemotherapy according to the usual clinical and radiological criteria adopted by the patient's attending physician.
  Interventions: Other: Usual clinical and radiological criteria

INTERVENTIONS:
Biological: Blood sampling — 20ml of patient peripherical blood will be collected
  Arms: Circulating Tumor Cells
Other: Usual clinical and radiological criteria — Clinical examination, tumoral evaluation
  Arms: Clinical and radiological criteria

SUMMARY:
Evaluation of the use of Circulating tumour Cells to guide chemotherapy from the 3rd line of chemotherapy for metastatic breast cancer.

DETAILED DESCRIPTION:
Phase III multicentre, randomized, open-label study comparing early evaluation of the efficacy of chemotherapy by determination of circulating tumour cells versus conventional clinical and radiological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 years.
* WHO performance status: 0 to 4.
* Metastatic breast cancer.
* Progression after 2 lines of chemotherapy with decision to initiate third-line chemotherapy.
* Disease evaluable by CTC (CTC-positive before starting chemotherapy).
* Histology: lobular or ductal adenocarcinoma.
* Information of the patient and signature of the informed consent form by the patient or her legal representative.

Exclusion Criteria:

* Disease not evaluable by CTC (CTC-negative before starting chemotherapy).
* History of other potentially metastatic cancer (stage III or IV cancer) different from breast cancer.
* Histology other than lobular or ductal adenocarcinoma.
* Pregnant woman, women likely to become pregnant or nursing mothers.
* Persons deprived of their freedom or under guardianship.
* Women unable to comply with the medical follow-up of the study for geographical, social or mental reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2010-03-02 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 7 years
  Overall survival (from date of randomization

SECONDARY OUTCOMES:
Measure of safety and tolerability | 7 years
  A list of the most frequent toxicity was established. The ranks 3 and 4 will be more specificaly collected.
Improvement of quality of life | 7 years
Time to progression, to discontinuation of therapy after 3rd line. | 7 years
Comparison of CTC with usual serum tumour markers | 7 years
Medico-economical analysis | 5 years
Estimate the clinical interest, in particular forecast, of the circulating tumoral DNA | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: PIERGA Jean-Yves, MD, Principal Investigator — Institut Curie
Locations (7):
- France (7):
  - Centre Georges Francois Leclerc, Dijon
  - Clinique Victor Hugo, Le Mans
  - Chu Limoges, Limoges
  - Institut Curie, Paris
  - Hopital Saint Louis, Paris
  - Institut Rene Huguenin Curie, Saint-Cloud
  - Institut de Canacerologie de L'Ouest, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabel L, Berger F, Cottu P, Loirat D, Rampanou A, Brain E, Cyrille S, Bourgeois H, Kiavue N, Deluche E, Ladoire S, Campone M, Pierga JY, Bidard FC. Clinical utility of circulating tumour cell-based monitoring of late-line chemotherapy for metastatic breast cancer: the randomised CirCe01 trial. Br J Cancer. 2021 Mar;124(7):1207-1213. doi: 10.1038/s41416-020-01227-3. Epub 2021 Jan 21. PMID 33473163
- [Result] Helissey C, Berger F, Cottu P, Dieras V, Mignot L, Servois V, Bouleuc C, Asselain B, Pelissier S, Vaucher I, Pierga JY, Bidard FC. Circulating tumor cell thresholds and survival scores in advanced metastatic breast cancer: the observational step of the CirCe01 phase III trial. Cancer Lett. 2015 May 1;360(2):213-8. doi: 10.1016/j.canlet.2015.02.010. Epub 2015 Feb 17. PMID 25700777